CLINICAL TRIAL: NCT01267006
Title: A Randomized Cross-over Study to Evaluate the Pharmacokinetics and Pharmacodynamics of Twice Daily Oral Administration of GSK1325756, Compared to Placebo, in Healthy Subjects; and the Pharmacokinetic Profile of Twice Daily Oral Administration of GSK1325756 in Healthy Fed and Fasted Elderly Subjects
Brief Title: Blood Levels and Effects of GSK1325756 in Healthy Adult Volunteers Aged 40 to 80 Years Old
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 114922
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — danirixin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Part A - Cohort 1 subjects will be administered GSK1325756 matching placebo tablets twice daily following a light meal for one day in accordance with the randomization schedule.
  Interventions: Drug: Placebo tablet
- GSK1325756 200 mg (Experimental): Part A - Cohort 1 subjects will be administered GSK1325756 200 mg immediate release tablets twice daily following a light meal for one day in accordance with the randomization schedule.
  Interventions: Drug: GSK1325756
- GSK1325756 50 mg (Experimental): Part A - Cohort 1 subjects will be administered GSK1325756 50 mg immediate release tablets twice daily following a light meal for one day in accordance with the randomization schedule.
  Interventions: Drug: GSK1325756
- GSK1325756 100 mg (Experimental): Part B - Cohort 2 subjects will be administered GSK1325756 100 mg following a light meal (Fed) or in the fasted state twice daily for one day in accordance with the randomization schedule.
  Interventions: Drug: GSK1325756

INTERVENTIONS:
Drug: GSK1325756 — GSK1325756 will be available as white, film coated immediate release tablets with dose strengths of 50 mg, 100 mg and 200 mg. The tablets will be administered twice daily by oral route with 240 milliliters of water.
  Arms: GSK1325756 100 mg; GSK1325756 200 mg; GSK1325756 50 mg
Drug: Placebo tablet — Placebo will be available as white film coated GSK1325756 matching tablet which will be administered twice daily by oral route with 240 milliliters of water.
  Arms: Placebo

SUMMARY:
This study will invite two groups of volunteers to participate.

The data from one group of volunteers will be used to find out how much study drug, known as GSK1325756, is in the blood after taking the drug twice in one day. Data will also collected to find out if the level of cetain blood cells, known as neutrophils, change significantly after taking the study drug twice in one day. This group of volunteers will be aged 40 to 64 years of age.

The data from the other group of volunteers will be used to find out if taking the study drug, GSK1325756, twice in one day with or without food, makes a difference to the level of study drug in the blood. This group of volunteers will also provide data to find out if any study drug metabolites are present in the bile, a fluid secreted by the liver. This group of volunteers will be aged 65 to 80 years of age.

DETAILED DESCRIPTION:
The current study will be conducted in two parts. In Part A - Cohort 1, healthy fed subjects aged 40 to 64 years (inclusive) will be enrolled to evaluate both the pharmacokinetics and pharmacodynamics of twice daily oral administration of GSK1325756 compared to matching placebo. In Part B - Cohort 2, healthy elderly subjects aged 65 to 80 years (inclusive) will be enrolled to evaluate the pharmacokinetic profile of twice daily oral administration of GSK1325756 for administered under fed and fasted conditions. Parts A and B may be performed in parallel.

The approximate duration of the current study is expected to be between 64 and 74 days. The study will require subjects to complete a screening visit within 30 days, followed by Part A - Cohort 1 enrolment requiring 3 x (3 day treatment period + 7 day washout period) or Part B Cohort 2 enrolment requiring 2 x (3 day treatment period + 7 day washout period). All subjects will complete a follow up visit within seven to 14 days of last dose.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-childbearing potential female who, at the at the time of signing the informed consent, aged between 40 and 64 years (inclusive) for enrolment in Part A - Cohort 1; between 65 and 80 years (inclusive) for enrolment in Part B - Cohort 2. A female of non-childbearing potential is defined as a pre-menopausal female with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<147 pmol/L) is confirmatory].
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures and objectives.
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase and bilirubin less than or equal to 1.5x Upper Limit of Normal (ULN) (isolated bilirubin greater than 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin less than 35%).
* Resting blood pressure (BP) of less than or equal to 140/90, irrespective of anti-hypertensive medication status for the subject.
* Body weight greater or equal to 60 kg for men and greater or equal to 45 kg for women; and Body Mass Index (BMI) within the range 19 to 32 kilograms per metres squared (kg/m2) (inclusive).
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study medication until one week post last dose.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A neutrophil count at screening of less than 2 x 10*9L. Repeat testing is not permitted.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive pre-study drug/alcohol screen, with the exception of a positive result considered by the investigator to be directly attributable to prescription medication approved for subject use during the study.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of greater than 21 units for males or greater than 14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
* Positive serum or urine human chorionic gonadotropin (hCG) test at screening or prior to first dose.
* Screening QT duration corrected for heart rate by Bazett's formula (QTcB) or QT correction for heart rate by Fridericia's formula (QTcF) greater than 450 msec; PR interval outside the range 120 to 200 msec or an ECG that it not suitable for QT measurements (e.g. poorly defined termination of T-wave).
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 3-months, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety, such as a subject who is taking a stable dose of anti-hypertensive medication for at least 3 months prior to the screening visit; or lipid lowering medications (statins or fibrates) for at least 3 months prior to the screening visit.
* Treatment with intravenous or intra-articular corticosteroids within 6 weeks of first dose of study medication.
* Current treatment with proton pump inhibitors (e.g. omeprazole, lansoprazole).
* Current treatment with H2-receptor antagonists (e.g. ranitidine or cimetidine).
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 3-month period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* Urinary cotinine or exhaled breath carbon monoxide (CO) levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.
* Direct involvement in the conduct of the study, or relative or any person directly involved in the conduct of the study

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-11-05 (Actual); Primary Completion 2011-01-27 (Actual); Study Completion 2011-01-27 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | 48 hours

SECONDARY OUTCOMES:
Pharmacodynamics | 48 hours
Adverse Events | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Bloomer JC, Nash M, Webb A, Miller BE, Lazaar AL, Beaumont C, Guiney WJ. Assessment of potential drug interactions by characterization of human drug metabolism pathways using non-invasive bile sampling. Br J Clin Pharmacol. 2013 Feb;75(2):488-96. doi: 10.1111/j.1365-2125.2012.04352.x. PMID 22670830
- See also: Results for study 114922 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114922?search=study&search_terms=114922#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 114922 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114922 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114922 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114922 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114922 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114922 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114922 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register